CLINICAL TRIAL: NCT01763970
Title: A Phase II Study of Hyperfractionated Stereotactic Radiotherapy in the Treatment of Metastatic Pediatric Sarcomas of Bony Sites
Brief Title: Stereotactic Radiation Therapy for Pediatric Sarcomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1367; NA_00070109 (Other: JHMIRB)
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Results first posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Sarcoma; Metastatic Disease; Bony Sites
Keywords: Stereotactic; Radiotherapy; Hypofractionated
MeSH Terms: conditions — Sarcoma; Neoplasm Metastasis | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hypofractionated SBRT (Experimental): 800 cGy delivered in 5 fractions every day to total dose of 4000 cGy
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT
  Other Names: Stereotactic Body Radiation Therapy (SBRT)

SUMMARY:
The stereotactic body radiation therapy (SBRT) literature focuses on clinical outcomes in the adult population. However, SBRT has a particularly strong rationale for application in pediatrics given that high biologically effective doses have been shown to increase control in histologies, such as sarcoma, which are common in the pediatrics population. With stereotactic radiation therapy techniques, a reduction in normal tissue dose surrounding the target lesion of interest may also be accomplished resulting in lower toxicity. Given that pediatric patients with sarcomas, presenting with limited metastases in lung and bone, are still considered to be a curable population with aggressive local therapy, SBRT could have a significant impact on outcomes in oligometastatic patients who may be otherwise unresectable.

DETAILED DESCRIPTION:
Pediatric patients with sarcoma who have limited metastases are still potentially curable with aggressive local therapy. However, conventional moderate dose radiation is unlikely to provide durable local control. Given the recent technologic advances in radiation delivery, it is now possible to deliver tumoricidal doses, using stereotactic radiation over a short time course with highly focal techniques. Stereotactic radiation has proven efficacious in the intracranial setting and in multiple extracranial sites in adults. It has not yet been well studied in the pediatrics population where there is a particularly strong rationale due to the ablative doses that can be delivered to tumor while simultaneously reducing high dose to normal tissues. The proposed trial is a single arm phase II study to determine the efficacy of SBRT in pediatric sarcomas with surgically unresectable metastatic disease. Oligometastatic sites eligible for treatment in this study include bony sites of disease. SBRT will be delivered to each eligible site to a total dose of 4000 delivered in 5 fractions of 800 per fractions each day. Following completion of SBRT, patients will undergo treatment response assessment with the use of diagnostic imaging, clinical examination, and completion of the Brief Pain Inventory to assess quality of life. The primary objective of this study is to determine the efficacy of SBRT delivered to a dose of 4000 centigray (cGy) in 5 fractions of 800 cGy each for patients greater than 3 years of age and < 40 years of age with metastatic disease of bone secondary to pediatric sarcoma. The secondary objectives of this study include describing the toxicity of SBRT with this regimen; assessing clinical response rate of each target lesion; assessing long-term clinical outcomes; and assessing quality of life following completion of treatment. For patients with potentially curable oligometastatic disease, surgical resection in conjunction with systemic therapy remains the standard of care. Patients on this study will continue to receive chemotherapy outside of the 2 week window for SBRT. Issues that may limit participation include our inability to assess late effects that may not develop till at least 10 years after therapy. For this reason, we will limit the population in this study to patients who are surgically unresectable and would be otherwise incurable with current standard systemic therapies.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed metastatic sarcoma of the soft tissue or bone
* must have measurable disease
* disease must be surgically unresectable as determined by a tumor board or surgeon
* greater than 3 years of age
* less than or equal to 40 years of age
* life expectancy of at least 9 months
* adequate performance status (Lansky Performance Status greater than or equal to 50).
* ability to understand and willingness to sign informed consent document

Exclusion Criteria:

* patients who have had chemotherapy or radiotherapy within 2 weeks prior to entering the study
* patients who have had any prior radiotherapy to the treatment site(s)
* patients may not participate on any other treatment protocol while they are receiving treatment on this protocol and for up to 3 months after these protocol treatments have ended
* pregnant women
* refusal of women of child bearing potential to take a pregnancy test prior to treatment

Ages: 4 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2020-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Ladra, M.D., Principal Investigator — The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (5):
- United States (5):
  - Stanford Medical Center, Stanford, California
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - St. Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Hypofractionated SBRT: This is a single-arm, prospective trial to examine the efficacy and safety of SBRT (SBRT) for the treatment of bone metastases in pediatric and young adult patients. Patients with metastatic nonrhabdomyosarcoma with bone metastases were treated with SBRT to a total dose of 40 Gy in 5 fractions (8 Gy/fraction). Physicians were permitted to treat up to five distinct lesions per patient.
Period: Overall Study
Arm/Group | Hypofractionated SBRT
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Hypofractionated SBRT: 800 delivered in 5 fractions every day to total dose of 4000
  SBRT: 800 delivered in 5 fractions every day to total dose of 4000
Arm/Group | Hypofractionated SBRT
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 17 [4 to 25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 9
  Non-Caucasian | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14
Lansky Play-Performance Scale (LPS) for Pediatric Functional Status [Count of Participants; unit: Participants] — The LPS for Pediatric Functional Status uses parent description of child's activity. A score of:
  100 - fully active 90 - minor restrictions in strenuous physical activity 80 - active, but gets tired more quickly 70 - greater restriction of play and less time spent in play activity 60 - up and around, but active play minimal 50 - lying around much of the day, but gets dressed 40 - mainly in bed; participates in quiet activities 30 - bedbound; needing assistance even for quiet play 20 - sleeping often; play entirely limited to very passive activities 10 - doesn't play 0 - unresponsive
  Participants
    LPS = 100 | 3
    LPS = 80-90 | 10
    LPS = 70 | 1
    LPS < 70 | 0
Histological type of cancer [Count of Participants; unit: Participants]
  Ewing sarcoma | 7
  Osteosarcoma | 3
  Soft-tissue sarcoma | 4
Number of Lesions Treated in Each Patient [Median (Full Range); unit: lesions] | 2.5 [1 to 5]
Consolidation of Metastatic Disease [Count of Participants; unit: Participants] — If a patient had all known sites of metastatic disease treated they were coded as total consolidation. If not all sites of metastatic disease were treated, they were coded as partial consolidation.
  Participants
    Total | 8
    Partial | 6
Prior systemic therapy [Count of Participants; unit: Participants] — Number of participants who received prior systemic therapy
  Participants | 14
Pain at baseline [Count of Participants; unit: Participants]
  Yes, has pain | 6
  No pain | 8
Treatment Duration [Median (Full Range); unit: days] | 7 [5 to 15]

OUTCOME MEASURES:

1. Primary Outcome: Lesion-specific Local Control at 6 Months Post-SBRT as Assessed by Percentage of Lesions Locally Controlled
Description: Local control was defined as the absence of local progression. Local progression was defined as:
  * (1) the development of a new soft tissue mass ≥1 cm at a site without a soft tissue component or with a soft tissue component <1 cm in at baseline
  * (2) an increase in the largest axial dimension of the soft tissue component by >20% in lesions with a ≥ 1 cm in soft tissue component at baseline
  * (3) a previous bone metastasis that was avid on fluorodeoxyglucose (FDG)-positron emission tomography (PET), became non-avid after SBRT, and then became avid again.
  The Kaplan-Meier method was used.
Time Frame: 6 months post-SBRT
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: lesions
Groups:
- Hypofractionated SBRT: SBRT: 800 centigray (cGy) delivered in 5 fractions every day to total dose of 4000 cGy
Arm/Group | Hypofractionated SBRT
Number analyzed (Participants) | 14
Number analyzed (lesions) | 37
percentage of lesions | 95 [68 to 99]

2. Secondary Outcome: Patient-specific Local Control at 6 Months Post-SBRT as Assessed by the Percentage of Patients Locally Controlled
Description: Patient-specific local control was calculated using the Kaplan-Meier method from initiation of SBRT to time of local failure. Patients who did not experience local failure were censored at the time of last follow up.
Time Frame: 6 months post-SBRT
Measure: Number (99% Confidence Interval); unit: percentage of patients
Groups:
- Hypofractionated SBRT: SBRT: 800 cGy delivered in 5 fractions every day to total dose of 4000 cGy
Arm/Group | Hypofractionated SBRT
Number analyzed (Participants) | 14
percentage of patients | 89 [43 to 98]

3. Secondary Outcome: Percentage of Patients With Progression-free Survival at 6 Months Post-SBRT
Description: To assess long-term clinical outcomes of this patient population after completion of SBRT by measuring progression-free survival. The Kaplan-Meier method was used to determine progression-free for survival from initiation of SBRT to progression (local or distant) or death due to any cause. Patients that did not have evidence of progression or who did not die, where censored at the time of last follow up.
Time Frame: 6 months post-SBRT
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Hypofractionated SBRT
Number analyzed (Participants) | 14
percentage of patients | 50 [23 to 93]

4. Secondary Outcome: Percentage of Patients With Overall Survival at 6 Months Post-SBRT
Description: The Kaplan-Meier method was used to calculate overall survival from initiation of SBRT to death due to any cause. Patients who had not died at the time of the analysis were censored at the time of last follow up.
Time Frame: 6 months post-SBRT
Measure: Number; unit: percentage of patients
Arm/Group | Hypofractionated SBRT
Number analyzed (Participants) | 14
percentage of patients | 100

5. Secondary Outcome: Change in Quality of Life (QoL) as Assessed by the Brief Pain Inventory
Description: Quality of life was assessed using the Brief Pain Inventory (BPI) form which assesses the severity of pain and impact on functioning on an 11-point scale at each follow up visit. Paired sample Wilcoxon signed-rank tests were performed to assess changes in pain scores on the Brief Pain Inventory; 0 being no pain and 10 being the worst pain.
Time Frame: Baseline and one-month post-SBRT
Population: BPI forms were completed for 10 patients at baseline and one-month post-SBRT.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hypofractionated SBRT
Number analyzed (Participants) | 10
score on a scale
  Baseline | 2 (2.4)
  One month | 2.1 (2.8)

6. Secondary Outcome: Number of Participants Experiencing Toxicity of SBRT
Description: To describe the toxicity of SBRT delivered to study patients measured by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Time Frame: 12 months after treatment starts
Measure: Count of Participants; unit: Participants
Arm/Group | Hypofractionated SBRT
Number analyzed (Participants) | 14
Participants | 9

7. Post Hoc Outcome: Progression-Free Survival by Consolidation Status
Description: The Kaplan-Meier method was used to calculate progression-free survival (in months) stratified by consolidation status (total consolidation vs. partial consolidation) from initiation of SBRT to progression (local or distant) or death due to any cause.
Time Frame: 3 years post-SBRT
Measure: Median (Inter-Quartile Range); unit: months
Groups:
- Partial Consolidation: SBRT: 800 cGy delivered in 5 fractions every day to total dose of 4000 cGy. Not all sites of metastatic disease were treated (partial consolidation).
- Total Consolidation: SBRT: 800 cGy delivered in 5 fractions to a total dose of 4000 cGy. All known sites of metastatic disease were treated.
Arm/Group | Partial Consolidation | Total Consolidation
Number analyzed (Participants) | 6 | 8
months | 3.7 [1.4 to 6.4] | 9.3 [3.0 to NA] — Upper limit not reached.

8. Post Hoc Outcome: Overall Survival by Consolidation Status
Description: The Kaplan-Meier method was used to calculate overall survival (in months) stratified by consolidation status (total consolidation vs. partial consolidation) from initiation of SBRT to death due to any cause.
Time Frame: 3 years post-SBRT
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Partial Consolidation | Total Consolidation
Number analyzed (Participants) | 6 | 8
months | 12.7 [9.8 to 24.2] | NA [23.3 to NA] — Median and upper limit not reached.

ADVERSE EVENTS:
Time Frame: 36 months.
Description: All of the adverse events were collected on systematic assessment except for the single patient who developed two grade 3 toxicities after treatment with SBRT. This patient developed osteonecrosis of the soft tissue of the wrist requiring curettage and grafting and subsequently fractured at the site of the graft. As such, this patient presented acutely and these toxicities were not picked up on systematic assessment.
Arm/Group | Hypofractionated SBRT
All-Cause Mortality (participants affected / at risk) | 8/14
Serious Adverse Events (participants affected / at risk) | 2/14
Other Adverse Events (participants affected / at risk) | 8/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypofractionated SBRT (N=14)
Esophagitis (Gastrointestinal disorders) | 1 (1) — CTCAE grade 3 esophagitis
Soft tissue necrosis and fracture (Musculoskeletal and connective tissue disorders) | 1 (2) — Necrosis of the distal radius requiring curettage and bone grafting approximately 22 months post-SBRT. The patient subsequently developed a fracture requiring operative repair at the bone graft site approximately 35 months post-SBRT.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypofractionated SBRT (N=14)
alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
myositis (Musculoskeletal and connective tissue disorders) | 1
Fatigue (General disorders) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Lower Extremity Weakness (Nervous system disorders) | 1 (1)
Wrist Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Compression Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Asymptomatic, grade 1
Paresthesia of the lower extremity (Nervous system disorders) | 1 (1) — Grade 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-21): https://cdn.clinicaltrials.gov/large-docs/70/NCT01763970/Prot_SAP_000.pdf